CLINICAL TRIAL: NCT04799574
Title: National Taipei University of Nursing and Health Sciences
Brief Title: Effect of Music Therapy in Improving the Physical Fitness and Depression in the Frailty of the Community Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, MEI - LING LU, Postgraduate of Master Degree, RN., National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ChenLu
Record Dates: First submitted 2020-06-07; First posted 2021-03-16 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Music Therapy; Frailty; Physical Fitness; Depression
Keywords: music therapy; frailty; physical fitness; depression; activity
MeSH Terms: conditions — Frailty; Depression; Motor Activity

STUDY DESIGN:
Intervention Model Description: one Experimental group and one Control group
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers in this study are the leaders of the activities and the nurses who had completed training in music therapy courses, and had obtained leadership certificates and qualifications in senior music activities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- music therapy activity (Experimental): The music therapy activity course design has a fixed process. The 90-minute course includes 10-15 minutes of warm-up activities, 50-60 minutes of main activities, 10-15 minutes of recovery activities, and 10 minutes of rest for the elders in the middle.
  Interventions: Other: music therapy activities
- Health education lecture (Placebo Comparator): routine activities of community
  Interventions: Other: music therapy activities

INTERVENTIONS:
Other: music therapy activities — Music therapy activity course design (Protocol):
  The researchers in this study are the leaders of the activities and the nurses who had completed training in music therapy courses and obtained a senior music activity leadership certificate and qualification, such as books and internship certificates. The course design uses the percussion music theory and Dalcroze and Orpff music pedagogy to plan activities, as follows:
  Each class in the music therapy activity course design has a fixed process. The 90-minute course includes 10-15 minutes of warm-up activities, 50-60 minutes of main activities, 10-15 minutes of recovery activities, and 10 minutes of rest for the elders in the middle. The content of the weekly main activities uses different music, musical instruments, props, or rhythms to lead the rhythm music activities.

SUMMARY:
Research Design This study adopted randomized clinical trials design, with two groups of pre-tests and post-tests, a single-blind test, a single-blind test, and intentional sampling. Four well-organized community care centers with the proper number of elderly people and the willingness to participate in Taipei City were selected to carry out the pre-test to screen out the qualified research subjects, and then, they were randomly assigned to the experimental group or control group. The experimental group received music therapy and routine activities, while the control group only received routine activities, and the researchers were the leaders of the music therapy activities. Data collection and fitness testing were performed by trained, certified, and qualified personnel. Before program implementation, a consensus meeting on testing consistency was conducted for the testers to obtain consistency in testing technology and scale questionnaires. The researchers were not involved in the testing, in order to ensure the independent position and blindness of the fitness testers. The study intervention was conducted for 12 weeks, once a week, 90 minutes each time. In the 13th week, the two groups performed the first post-test, while the second post-test was in the 16th week.

Research Structure The independent variables include demographic data, and one or more of the five indicators of disease state and physical status decline. The intervention measures include various music therapy activities, and the dependent variables are the performance indicators including: frailty indicators (BMI, grip strength, 2.44 meters of timed get-up-and-go, 30 seconds of sit-to-stand, 2 minutes of knee bending and leg raising), physical activity, conscious health status, and depression. This study explores the effectiveness of music therapy in improving the physical fitness, degree of activity, and depression of elderly in the community.

DETAILED DESCRIPTION:
Music therapy activity course design (Protocol):

The researchers in this study are the leaders of the activities and the nurses who had completed training in music therapy courses and obtained a senior music activity leadership certificate and qualification, such as books and internship certificates. The course design uses the percussion music theory and Dalcroze and Orpff music pedagogy to plan activities, as follows:

Each class in the music therapy activity course design has a fixed process. The 90-minute course includes 10-15 minutes of warm-up activities, 50-60 minutes of main activities, 10-15 minutes of recovery activities, and 10 minutes of rest for the elders in the middle. The content of the weekly main activities uses different music, musical instruments, props, or rhythms to lead the rhythm music activities.

Research Subjects:

1. The case acceptance conditions of this study are as follows:

The case should be at least 65 years old. The case should meet one or more of Fried Frailty's 5 screening conditions or have a depression index ≥ 15 points.

The case should be capable of language expression and freedom of movement. 2. The exclusion conditions are as follows:

(1). Those who do not meet the frailty condition and depression tendency (2). Those who cannot participate in the study in the scheduled time. (3). Those with difficulty in language expression and mobility. Research Structure The independent variables include demographic data, and one or more of the five indicators of disease state and physical status decline. The intervention measures are various activities of music therapy, and the dependent variables are the performance indicators including: frailty indicators (BMI, grip strength, 2.44 meters of time get-up-and-go, 30 seconds of sit-to-stand, 2 minutes of knee bending and leg raising), physical activity, conscious health status and depression. Explore the effectiveness of music therapy in improving the physical fitness, activity and depression of the elderly in the community.

Definition of terms and use of tools

Demographic variables refer to:

The basic data of the research subjects including 8 items such as age, gender, education level, marital status, living situation, economic source, economic status, and food preparation methods.

The disease state refers to:

Study the physical health status of the research subjects, including types of chronic diseases, types of drugs taken daily, conscious health status and emotional status.

Music therapy:

It refers to the music activities led by the medical staff who had completed training in music therapy courses during the entire research program, with the curriculum designed to suit the health needs of the elder group. The researchers in this study are the leaders of the activities and also the nurses who had completed training in music therapy courses and obtained a senior music activity leadership certificate and qualifications such as books and internship certificates. The course design uses percussion music theory and Dalcroze and Orpff music pedagogy to plan activities.

Physical fitness:

The physical fitness in this study mainly includes cardiopulmonary endurance, muscle power, and body mass index. Muscle power test measures the grip strength of the dominant hand and lower limb muscle power. This study uses Smedlay Dynamometer 100Kg YOII model grip strength meter, its retest reliability is based on the highest retest reliability using the average of 2 rounds of the intraclass correlation coefficient (ICC) (ICC = 0.88). This study is based on the Fried Frailty Standard, and the grip strength of the dominant hand is calculated by the BMI of the elderly. Lower extremity muscle power is the ability to assess the individual's movement capacity and is tested with the "30-second sit-to-stand" test in Senior Fitness Test (SFT) published by Rikil and Jones in 1999 to mainly access the lower extremity muscle power and daily life movement capacity of the elderly. The physical fitness of the elderly in this study is determined by the Health Promotion Administration fitness test. The normal value of "30-second sit-and-stand" should be greater than 12 times for men and 10 times for women; cardiopulmonary endurance is measured by "2.44 meters of time get-up-and-go" and "2-minute knee bending and leg raising". The norm of men and women's "2.44 meters of time get-up-and-go" in Taiwan is ≦ 8 seconds or walking speed <0.8 meters/second "2-minute knee bending and leg raising" is an indicator of the endurance of systemic exercise. The normal value is more than 90 times for men and more than 80 times for women.

Activity:

In this study, the activity test scale-International Physical Activity Questionnaire-Self-filled short version of Taiwan Chinese version, International Physical Activity Questionnaire (IPAQ-SF) translated and developed by Professor Liu Yingmei in cooperation with Ministry of Health and Welfare was adopted. In the self-filled Chinese version, the English and Chinese language conformity, and the content validity index of similarity of meaning are .994, and .992; the intrinsic level correlation coefficient of the Chinese and English versions is .704, which has good reliability and validity as well as cultural sensitivity.

Depression:

This study uses the Taiwan Geriatric Depression Scale (TGDS-30). The scale has a total of 30 questions. The question is answered based on the condition of the last week. It can be self-filled or structured. The answer is dichotomous (yes/no), with a total score of 0-30 points. A total score of more than 15 points means one is suspected of suffering from depression. A higher score indicates a higher degree of depression. Therefore, the standard for accepting cases in this study is TGDS-30 depression index ≥ 15 points. In terms of reliability of this scale, the Cronbachα value of the overall scale is 0.94, the retest reliability is 0.82, and the halving reliability is 0.95; in terms of validity, the validity and reliability have 93.3% sensitivity and 92.3% specificity, so it is a test scale with good reliability and validity.

Frailty:

It refers to the Health Promotion Administration Assessment Standards for Physical Fitness of the Elderly and the criteria for five indicators of frailty proposed by Fried in 2001 for the indicators of frailty. Failure to meet any of the indicators means no frailty, meeting one or two indicators are pre-frailty, and meeting three or more indicators are frailty.

This study accepts the case who meets one or more indicators.

Conscious health status:

The researcher draws a 10 cm straight line on the white paper, with 1 marked on the left end and 10 on the right end, explains the meaning of 1 and 10 to the elders, and asks the elders to point out the conscious health status on the line. Then the researcher measures the score with a ruler, and the data is calculated to the first decimal point. From 1-10, 1 means poor conscious health, 10 means very good conscious health, and ≦ 5 cm or less means that the conscious health status is not good.

ELIGIBILITY:
Inclusion Criteria:

1. Should be at least 65 years old.
2. Should meet one or more of the 5 screening conditions of the Fried Frailty Scale or have a depression index ≥ 15 points.
3. Should be capable of language expression and freedom of movement.

Exclusion Criteria:

1. . Those who do not meet the frailty condition or depression tendency
2. . Those who cannot participate in the study in the scheduled time.
3. . Those with difficulty in language expression and mobility.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-05-27 (Actual)

PRIMARY OUTCOMES:
Depression index | 0 weeks(pre-test)
  This study uses the Taiwan Geriatric Depression Scale (TGDS-30), which has a total of 30 questions. The answers are dichotomous (yes/no), and are scored between 0-30 points, where a total score of more than 15 points means one is suspected of suffering from depression, and a higher score indicates a higher degree of depression.
Depression index | 1 week after the 12-week intervention is completed (post-test 1)
  This study uses the Taiwan Geriatric Depression Scale (TGDS-30), which has a total of 30 questions. The answers are dichotomous (yes/no), and are scored between 0-30 points, where a total score of more than 15 points means one is suspected of suffering from depression, and a higher score indicates a higher degree of depression.
Depression index | 4 weeks after the 12-week intervention is completed (post-test 2)
  This study uses the Taiwan Geriatric Depression Scale (TGDS-30), which has a total of 30 questions. The answers are dichotomous (yes/no), and are scored between 0-30 points, where a total score of more than 15 points means one is suspected of suffering from depression, and a higher score indicates a higher degree of depression.
The International Physical Activity Questionnaire Short Form (IPAQ-SF) | 0 weeks(pre-test)
  This study adopted the Taiwanese Chinese version of the activity test scale of the International Physical Activity Questionnaire-Self-filled short version (IPAQ-SF), as translated and developed by Professor Liu Ying Mei in cooperation with the Ministry of Health and Welfare. The contents of the self-filled Chinese version conform to create valid content with meanings similar to the English version, .994, and .992, respectively. The intrinsic level of the correlation coefficient of the Chinese and English versions is .704, which has good reliability and validity, as well as cultural sensitivity. The IPAQ short version includes walking (W), medium-intensity activity (M), high-intensity activity (V), and overall physical activity scores. All consecutive scores are expressed in METs-minutes/week. Walking=3.3METS, medium-intensity activity=4.0METS, high-intensity activity=8.0METSThe higher the score, the higher the level of participation in the activity.
The International Physical Activity Questionnaire Short Form (IPAQ-SF) | 1 week after the 12-week intervention is completed (post-test 1)
  This study adopted the Taiwanese Chinese version of the activity test scale of the International Physical Activity Questionnaire-Self-filled short version (IPAQ-SF), as translated and developed by Professor Liu Ying Mei in cooperation with the Ministry of Health and Welfare. The contents of the self-filled Chinese version conform to create valid content with meanings similar to the English version, .994, and .992, respectively. The intrinsic level of the correlation coefficient of the Chinese and English versions is .704, which has good reliability and validity, as well as cultural sensitivity. The IPAQ short version includes walking (W), medium-intensity activity (M), high-intensity activity (V), and overall physical activity scores. All consecutive scores are expressed in METs-minutes/week. Walking=3.3METS, medium-intensity activity=4.0METS, high-intensity activity=8.0METSThe higher the score, the higher the level of participation in the activity.
The International Physical Activity Questionnaire Short Form (IPAQ-SF) | 4 weeks after the 12-week intervention is completed (post-test 2)
  This study adopted the Taiwanese Chinese version of the activity test scale of the International Physical Activity Questionnaire-Self-filled short version (IPAQ-SF), as translated and developed by Professor Liu Ying Mei in cooperation with the Ministry of Health and Welfare. The contents of the self-filled Chinese version conform to create valid content with meanings similar to the English version, .994, and .992, respectively. The intrinsic level of the correlation coefficient of the Chinese and English versions is .704, which has good reliability and validity, as well as cultural sensitivity. The IPAQ short version includes walking (W), medium-intensity activity (M), high-intensity activity (V), and overall physical activity scores. All consecutive scores are expressed in METs-minutes/week. Walking=3.3METS, medium-intensity activity=4.0METS, high-intensity activity=8.0METSThe higher the score, the higher the level of participation in the activity.

SECONDARY OUTCOMES:
physical fitness: 30-second sit-to-stand | 0 weeks(pre-test)
  "30-second sit-to-stand" test in the Senior Fitness Test (SFT), to mainly assess the lower extremity muscle power. The normal value of completing "30-second sit-and-stand" should be greater than 12 times for men and 10 times for women. The more times the better.
physical fitness: 30-second sit-to-stand | 1 week after the 12-week intervention is completed (post-test 1)
  "30-second sit-to-stand" test in the Senior Fitness Test (SFT), to mainly assess the lower extremity muscle power. The normal value of completing "30-second sit-and-stand" should be greater than 12 times for men and 10 times for women. The more times the better.
physical fitness: 30-second sit-to-stand | 4 weeks after the 12-week intervention is completed (post-test 2)
  "30-second sit-to-stand" test in the Senior Fitness Test (SFT), to mainly assess the lower extremity muscle power. The normal value of completing "30-second sit-and-stand" should be greater than 12 times for men and 10 times for women. The more times the better.
physical fitness: 2-minute knee bending and leg raising | 0 weeks(pre-test)
  "2-minute knee bending and leg raising", which is an indicator of endurance in systemic exercise, and the normal values are more than 90 times for men and more than 80 times for women. The more times the better.
physical fitness: 2-minute knee bending and leg raising | 1 week after the 12-week intervention is completed (post-test 1)
  "2-minute knee bending and leg raising", which is an indicator of endurance in systemic exercise, and the normal values are more than 90 times for men and more than 80 times for women. The more times the better.
physical fitness: 2-minute knee bending and leg raising | 4 weeks after the 12-week intervention is completed (post-test 2)
  "2-minute knee bending and leg raising", which is an indicator of endurance in systemic exercise, and the normal values are more than 90 times for men and more than 80 times for women. The more times the better.
physical fitness: 2.44 meters of timed get-up-and-go | 0 weeks(pre-test)
  "2.44 meters of timed get-up-and-go", where the norm for both men and women in Taiwan is ≦ 8 seconds or walking speed of <0.8 meters/second, The less time the better.
physical fitness: 2.44 meters of timed get-up-and-go | 1 week after the 12-week intervention is completed (post-test 1)
  "2.44 meters of timed get-up-and-go", where the norm for both men and women in Taiwan is ≦ 8 seconds or walking speed of <0.8 meters/second, The less time the better.
physical fitness: 2.44 meters of timed get-up-and-go | 4 weeks after the 12-week intervention is completed (post-test 2)
  "2.44 meters of timed get-up-and-go", where the norm for both men and women in Taiwan is ≦ 8 seconds or walking speed of <0.8 meters/second, The less time the better.
physical fitness: grip strength | 0 weeks(pre-test)
  This study uses the Smedlay Dynamometer 100Kg YOII grip strength meter, which is based on the highest retest reliability and uses the average of 2 rounds as the intraclass correlation coefficient (ICC) (ICC = 0.88). This study is based on the Fried Frailty Standard, and the grip strength of the dominant hand is calculated according to the BMI of the elderly.
physical fitness: grip strength | 1 week after the 12-week intervention is completed (post-test 1)
  This study uses the Smedlay Dynamometer 100Kg YOII grip strength meter, which is based on the highest retest reliability and uses the average of 2 rounds as the intraclass correlation coefficient (ICC) (ICC = 0.88). This study is based on the Fried Frailty Standard, and the grip strength of the dominant hand is calculated according to the BMI of the elderly.
physical fitness: grip strength | 4 weeks after the 12-week intervention is completed (post-test 2)
  This study uses the Smedlay Dynamometer 100Kg YOII grip strength meter, which is based on the highest retest reliability and uses the average of 2 rounds as the intraclass correlation coefficient (ICC) (ICC = 0.88). This study is based on the Fried Frailty Standard, and the grip strength of the dominant hand is calculated according to the BMI of the elderly.
Conscious health status 1-10 | 0 weeks(pre-test)
  The researcher drew a 10 cm straight line, with 1 marked on the left end and 10 on the right end, explained the 1 to 10 rating system to the elders, where 1 denotes poor conscious health, 10 denotes very good conscious health, and ≦ 5 cm or less denotes that the conscious health status is not good.
Conscious health status 1-10 | 1 week after the 12-week intervention is completed (post-test 1)
  The researcher drew a 10 cm straight line, with 1 marked on the left end and 10 on the right end, explained the 1 to 10 rating system to the elders, where 1 denotes poor conscious health, 10 denotes very good conscious health, and ≦ 5 cm or less denotes that the conscious health status is not good.
Conscious health status 1-10 | 4 weeks after the 12-week intervention is completed (post-test 2)
  The researcher drew a 10 cm straight line, with 1 marked on the left end and 10 on the right end, explained the 1 to 10 rating system to the elders, where 1 denotes poor conscious health, 10 denotes very good conscious health, and ≦ 5 cm or less denotes that the conscious health status is not good.

CONTACTS AND LOCATIONS:
Overall Officials: Miao Yen Chen, Ph.D., Study Director — National Taipei University of Nursing and Health Sciences
Locations (1):
- National Taipei University of Nursing and Health Sciences, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
After the article is published, the research data can be shared

REFERENCES:
- [Result] Drey M, Pfeifer K, Sieber CC, Bauer JM. The Fried frailty criteria as inclusion criteria for a randomized controlled trial: personal experience and literature review. Gerontology. 2011;57(1):11-8. doi: 10.1159/000313433. Epub 2010 Apr 21. PMID 20407227
- [Result] Mahendran R, Rawtaer I, Fam J, Wong J, Kumar AP, Gandhi M, Jing KX, Feng L, Kua EH. Art therapy and music reminiscence activity in the prevention of cognitive decline: study protocol for a randomized controlled trial. Trials. 2017 Jul 12;18(1):324. doi: 10.1186/s13063-017-2080-7. PMID 28701205
- [Result] Castaneda-Gameros D, Redwood S, Thompson JL. Physical Activity, Sedentary Time, and Frailty in Older Migrant Women From Ethnically Diverse Backgrounds: A Mixed-Methods Study. J Aging Phys Act. 2018 Apr 1;26(2):194-203. doi: 10.1123/japa.2016-0287. Epub 2018 Mar 23. PMID 28605284
- [Result] Dumitrache CG, Rubio L, Rubio-Herrera R. Perceived health status and life satisfaction in old age, and the moderating role of social support. Aging Ment Health. 2017 Jul;21(7):751-757. doi: 10.1080/13607863.2016.1156048. Epub 2016 Mar 8. PMID 26954480
- [Result] Vuilleumier P, Trost W. Music and emotions: from enchantment to entrainment. Ann N Y Acad Sci. 2015 Mar;1337:212-22. doi: 10.1111/nyas.12676. PMID 25773637
- [Result] Kim JH, Kim JM. Subjective life expectancy is a risk factor for perceived health status and mortality. Health Qual Life Outcomes. 2017 Oct 2;15(1):190. doi: 10.1186/s12955-017-0763-0. PMID 28969645
- [Result] Modig S, Midlov P, Kristensson J. Depressive symptoms among frail elderly in ordinary living: who is affected and who is treated? Aging Ment Health. 2014;18(8):1022-8. doi: 10.1080/13607863.2014.903469. Epub 2014 Apr 7. PMID 24708142
- [Result] Ishikawa M, Yamanaka G, Yamamoto N, Nakaoka T, Okumiya K, Matsubayashi K, Otsuka K, Sakura H. Depression and Altitude: Cross-Sectional Community-Based Study Among Elderly High-Altitude Residents in the Himalayan Regions. Cult Med Psychiatry. 2016 Mar;40(1):1-11. doi: 10.1007/s11013-015-9462-7. PMID 26162459
- [Result] Costa SN, Vieira ER, Bento PCB. Effects of Home- and Center-Based Exercise Programs on the Strength, Function, and Gait of Prefrail Older Women: A Randomized Control Trial. J Aging Phys Act. 2020 Jan 1;28(1):122-130. doi: 10.1123/japa.2018-0363. PMID 31629355
- [Result] Leiros-Rodriguez R, Soto-Rodriguez A, Perez-Ribao I, Garcia-Soidan JL. Comparisons of the Health Benefits of Strength Training, Aqua-Fitness, and Aerobic Exercise for the Elderly. Rehabil Res Pract. 2018 Jun 19;2018:5230971. doi: 10.1155/2018/5230971. eCollection 2018. PMID 30018825
- [Result] Lohne-Seiler H, Kolle E, Anderssen SA, Hansen BH. Musculoskeletal fitness and balance in older individuals (65-85 years) and its association with steps per day: a cross sectional study. BMC Geriatr. 2016 Jan 12;16:6. doi: 10.1186/s12877-016-0188-3. PMID 26755421